CLINICAL TRIAL: NCT04162431
Title: Diagnosis Of Lymphoma In Vivo Using Vibrational Spectroscopy (Ex Vivo Phase)
Brief Title: DOLPHIN-VIVO: Diagnosis Of LymPHoma IN Vivo (Ex Vivo Phase)
Acronym: DOLPHIN-VIVO
Status: Completed | Type: Observational
Sponsor: University of Exeter (Other)
Collaborators: Gloucestershire Hospitals NHS Foundation Trust (Other); University of Bristol (Other)
Responsible Party: Sponsor
Other Study IDs: 1819/31; 258155 (Registry Identifier: IRAS); II-LB-1117-20002 (Other Grant/Funding Number: NIHR)
Record Dates: First submitted 2019-11-11; First posted 2019-11-14 (Actual); Last update posted 2024-06-11 (Actual); Status verified 2024-06

CONDITIONS: Lymphoma; Head and Neck Cancer
Keywords: Raman; Lymphoma
MeSH Terms: conditions — Lymphoma; Head and Neck Neoplasms | interventions — Nonlinear Optical Microscopy; Biopsy, Fine-Needle; Cytological Techniques

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Bisected fresh frozen lymph nodes
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- non-hodgkin lymphoma: patients diagnosed with non-hodgkin lymphoma
  Interventions: Diagnostic Test: spectroscopic measurement; Diagnostic Test: FNA biopsy; Diagnostic Test: histopathology and cytology
- hodgkin lymphoma: patients diagnosed with hodgkin lymphoma
  Interventions: Diagnostic Test: spectroscopic measurement; Diagnostic Test: FNA biopsy; Diagnostic Test: histopathology and cytology
- squamous cell carcinoma: patients diagnosed with squamous cell carcinoma
  Interventions: Diagnostic Test: spectroscopic measurement; Diagnostic Test: FNA biopsy; Diagnostic Test: histopathology and cytology
- reactive: patients diagnosed with a reactive (non-cancerous) lymph node
  Interventions: Diagnostic Test: spectroscopic measurement; Diagnostic Test: FNA biopsy; Diagnostic Test: histopathology and cytology
- other: none of the above. Other cancer and non-cancer conditions
  Interventions: Diagnostic Test: spectroscopic measurement; Diagnostic Test: FNA biopsy; Diagnostic Test: histopathology and cytology

INTERVENTIONS:
Diagnostic Test: spectroscopic measurement — measurement of the tissue with spectroscopy
  Other Names: raman; infra red
Diagnostic Test: FNA biopsy — a fine needle aspiration (FNA) biopsy will be taken
  Other Names: fine needle aspiration biopsy
Diagnostic Test: histopathology and cytology — Histopathology and cytology will be performed on the samples

SUMMARY:
Lymphoma diagnosis often involves removal and biopsy of one or more lymph nodes. Many (around half) of these diagnostic procedures show that no cancer is present, hence unnecessary removal results in numerous side effects and complications. The procedure is also highly invasive.

The investigators have already shown that it is possible to tell the difference between healthy and diseased tissue in the laboratory by looking at the light emitted by tissue when a low power laser is shone on to it. The investigators intend to use this technique, known as "Raman Spectroscopy" (RS) to tell if tissue in the node is cancerous or healthy. By combining RS with a fine needle, the technique can target tissues below the skin with minimal invasion. Our needle will provide the clinician with instant diagnosis without the delay and cost of a laboratory analysis by pathologists.

The investigators have designed a probe that slides through a fine needle, guided by ultrasound, to the lymph node. The space between the two needles provides space for cell aspirate.

The investigators propose to measure spectra from excess lymph node biopsy samples taken during standard routine diagnostic biopsy.

The investigators are also interested to see if they can successfully extract a fine needle aspiration (FNA) biopsy sample using the device, as well as record a RS measurement. If successful this would ease clinical adoption as the study could run in parallel with existing standard routine clinical practice, using just one device.

This study will evaluate the new device on half a lymph node that will be excised and snap-frozen during a routine surgical biopsy, to gather data for submission of approvals for an in-vivo study to follow.

DETAILED DESCRIPTION:
Surplus lymph node tissue collected from patients undergoing routine surgical treatment for head & neck disease will be investigated using vibrational spectroscopy.

The project will develop a combined FNA/Raman spectroscopy needle probe. This study will evaluate this device on excised lymph node tissue to gather data for submission of approvals for an in-vivo study to follow. Raman & FTIR (fourier transform infrared) spectra will be correlated with routine histopathology results using multivariate analysis methods. Cytology samples taken using the device will be compared with histopathology results.

Aims

To demonstrate that the FNA/Raman spectroscopy probe device, developed as part of this project, can:

Safely perform measurement of Raman spectra on excised lymph node tissue Safely perform FNA (fine needle aspiration) biopsies on excised lymph node tissue To evaluate the performance of a Raman needle probe to detect lymphoma & malignancy in excised head & neck lymph nodes and differentiate from benign nodes.

To develop the investigators understanding of vibrational spectroscopy signal characteristics in head & neck lymph nodes (through Raman & FTIR mapping measurements of tissue sections).

Objectives To test a new combined FNA and spectroscopic device on ex vivo tissue in preparation for an in vivo study.

Outcome

Primary Outcome Measures The FNA/Raman spectroscopy probe device can be used safely on excised lymph nodes to measure tissue spectra and collect FNA biopsies.

Diagnostic performance of vibrational spectroscopy for differentiation of lymphoma & malignant nodes from benign nodes.

Secondary Outcome Measures Evaluation of the performance of a Raman needle probe to detect lymphoma & malignancy in excised head & neck lymph nodes and differentiate from benign nodes. To develop the investigators understanding of vibrational spectroscopy signal characteristics in head & neck lymph nodes (through Raman & FTIR mapping measurements of tissue sections).

Evaluation of the performance of a Raman needle probe to measure head & neck lymph nodes (ergonomic design, ease of use etc.).

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing biopsy or excision of lymph nodes as part of their routine clinical care within Gloucestershire Hospitals NHS Foundation Trust.
* Patients undergoing lymphadenectomy as part of routine treatment

Exclusion Criteria:

* Patients unable to consent to the study due to communication difficulties
* Patients unable to consent to the study due to lack of capacity

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients undergoing surgical head & neck lymph node biopsy within Gloucestershire Hospitals NHS Foundation Trust Patients with a lump in their head or neck are sometimes referred by their GP for a biopsy. This often first involves taking a small sample of cells with a fine needle, guided by ultrasound, called a Fine Needle Aspiration (FNA) biopsy. If the result from this FNA biopsy is inconclusive, then they are often further referred for a surgical biopsy. Gloucestershire Hospitals NHS Foundation Trust is a tertiary referral centre for surgical head and neck biopsies.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2021-06-28 (Actual); Primary Completion 2024-06-07 (Actual); Study Completion 2024-06-07 (Actual)

PRIMARY OUTCOMES:
Safe spectroscopic measurement | 3 years
  The FNA/Raman spectroscopy probe device can be used safely on excised lymph nodes to measure tissue spectra and collect FNA biopsies.
Diagnostic discrimination | 3 years
  Diagnostic performance of vibrational spectroscopy for differentiation of lymphoma & malignant nodes from benign nodes

SECONDARY OUTCOMES:
Cancer Performance evaluation | 3 years
  Evaluation of the performance of a Raman needle probe to detect lymphoma & malignancy in excised head & neck lymph nodes and differentiate from benign nodes
Understanding of Raman on lymph nodes | 3 years
  To develop our understanding of vibrational spectroscopy signal characteristics in head & neck lymph nodes (through Raman & FTIR mapping measurements of tissue sections).
General Performance evaluation | 3 years
  Evaluation of the performance of a Raman needle probe to measure head & neck lymph nodes (ergonomic design, ease of use etc.)

CONTACTS AND LOCATIONS:
Overall Officials: Nick Stone, Study Director — University of Exeter
Locations (1):
- Gloucestershire Hospitals NHS Foundation Trust, Gloucester, Gloucestershire, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Unique study number and MRN (medical records number) (hospital number)